CLINICAL TRIAL: NCT06122376
Title: Clinical Safety and Efficacy of AutoBrush® 360° U-Shaped Sonic Toothbrush on Plaque and Gingivitis in a 30-Day Model
Brief Title: Plaque and Gingivitis Evaluation of a U-Shaped Toothbrush in a 30-Day Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lander Enterprises, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AB-GBP-2023-02
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Plaque Induced Gingivitis
Keywords: gingivitis; dental plaque; Power toothbrush; manual toothbrush
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Examiner-blind only, subjects received treatment assignment and instructions in a room separate from the examiner and exam area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- U-shaped power toothbrush (Experimental): U-shaped power toothbrush with fluoride toothpaste
  Interventions: Device: U-shaped Power Toothbrush
- Manual Toothbrush (Placebo Comparator): soft manual toothbrush with fluoride toothpaste
  Interventions: Device: Soft Manual Toothbrush

INTERVENTIONS:
Device: U-shaped Power Toothbrush — Twice daily brushing for 30 seconds with fluoride toothpaste
  Arms: U-shaped power toothbrush
Device: Soft Manual Toothbrush — Twice daily brushing for two minutes with fluoride toothpaste
  Arms: Manual Toothbrush

SUMMARY:
The objective of this 30 day, randomized, two group, parallel, examiner-blind clinical trial is to assess the safety and efficacy of AutoBrush® 360° U-shaped Sonic Toothbrush on plaque and gingivitis, compared to an American Dental Association (ADA) reference manual soft toothbrush. The extent of gingival abrasion and recession and oral safety will be evaluated.

DETAILED DESCRIPTION:
This single-center, randomized, controlled, examiner-blind, 30-day parallel study will consist of Screening and Baseline visits with approximately 80 subjects (age 5-65 years) who will read and sign an informed consent form and assent form, assessed for evidence of gingivitis and plaque according to the Modified Gingival Index (MGI) and the Lobene-Soparkar Modification of Turesky Modified Quigley-Hein Plaque Index (LSPI) at Baseline, Day 15 and Day 30. Gingival recession and gingival abrasion will be measured at all visits. Subjects will be randomly assigned to one of two groups twice daily brushing with ADA accepted fluoride toothpaste and 1) two-minute brushing with ADA reference standard manual toothbrush, or 2) 30-second brushing with AutoBrush® 360° U-shaped Sonic Toothbrush.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy males and females at least 5 to 65 years of age.
* If under age 18, willing to provide assent to participate and consent from a parent or legal guardian prior to being entered into the study; If 18 years of age or older, is able to read, sign and receive a copy of the signed informed consent form.
* regular manual toothbrush users and able to brush their own teeth on a daily basis.
* In good health based on medical history review by the investigator.
* willing to refrain from all oral hygiene for approximately 12-16 hours prior to each study visit and discontinue eating and drinking for approximately 30 minutes prior to each study visit, with the exception of sips of water.
* Have a minimum of 18 natural teeth, in the adult dentition, with scorable facial and lingual surfaces. If under the age of 12, must have at least 12 fully erupted teeth, primary or permanent teeth. Partially erupted permanent teeth and primary teeth that are loose or in process of exfoliation will not be included in the tooth count. Teeth that are grossly carious, orthodontically banded, exhibiting general cervical abrasion and/or enamel abrasion, > 2 mm gingival recession will not be included in the tooth count.
* Present with a gingival index score ≥ 1.75 according to the Modified Gingival Index at Baseline, a plaque index score > 1.80 according to the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index, following a 12 to 16-hour plaque accumulation period at Baseline.
* willing and able to refrain from dental treatment during the course of the study, except on an emergency basis.

Exclusion Criteria:

* history of adverse effects, oral soft or hard tissue sensitivity, to any ingredient in the test materials.
* Self-reported serious medical conditions.
* Self-reported as pregnant or nursing.
* Under treatment for a heart condition requiring use of pacemaker.
* Have any condition, in the opinion of the investigator, that would place the subject at increased risk or preclude the subject's full compliance with or completion of the study?
* Require antibiotic premedication prior to dental procedures.
* Have had antibiotic, anti-inflammatory, anti-coagulant medication or chemotherapeutic antiplaque/antigingivitis therapy within 30 days of screening exams.
* participated in any study involving oral care products, concurrently or within the 30 days of screening exams.
* Unwilling to discontinue use of other oral hygiene products for the duration of the study.
* Present use of any tobacco products.
* Presence of severe periodontal disease or being actively treated for periodontal disease.
* Have grossly carious, fully crowned, or extensively restored teeth.
* Have orthodontic appliances, peri/oral piercings, or removable partial dentures.
* Have significant oral soft tissue pathology based on a visual examination.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Gingivitis: Modified Gingival Index | Whole mouth mean change from Baseline in MGI scores at Day 30.
  Gingival Inflammation, assessed on a 5-point scale (0 to 4), will be scored in six areas (disto-buccal, mid-buccal and mesio-buccal, disto-lingual, mid-lingual and mesio-lingual) of all scorable teeth using criteria: 0 = Normal (absence of inflammation), 1 = Mild inflammation (slight change in color, little change in texture) of any portion of the entire gingival unit; 2 = Mild inflammation of the entire gingival unit; 3 = Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit; 4 = Severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.
Plaque: Lobene-Soparkar Modification of Turesky Modification of Quigley-Hein Plaque Index | Whole mouth mean change in LSPI scores at Day 30, immediate post-brushing (Pre- to Post-Brushing scores)
  Plaque will be disclosed using a red disclosing solution and each tooth will be scored in six areas (disto-buccal, mid-buccal and mesio-buccal, disto-lingual, mid-lingual and mesio-lingual), according to the criteria noted below: 0 = No plaque; 1 = Separate flecks or discontinuous band of plaque at the gingival (cervical) margin; 2 = Thin (up to 1 mm), continuous band of plaque at the gingival margin; 3 = Band of plaque wider than 1 mm but less than 1/3 of tooth surface area; 4 = Plaque covering 1/3 or more, but less than 2/3 of tooth surface area; 5 = Plaque covering 2/3 or more of tooth surface area.

SECONDARY OUTCOMES:
Gingivitis | Change from Baseline at Day 15 and Day 30
  Whole mouth MGI, Gumline MGI, Proximal, Mean distal score of the last posterior tooth in each quadrant.
Plaque | Change from Baseline at Day 15 and Day 30
  LSPI: Whole mouth, Gumline, Proximal, distal score of the last posterior tooth in each quadrant.
Safety: gingival recession | Changes from Baseline at Day 15 and Day 30
  Gingival recession measurements (mm) will be carried out at six sites per tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual). Recession will be measured as the visible distance from the cemento-enamel junction (CEJ) to the gingival margin.
Safety: gingival abrasion | Changes from Baseline at Day 15 and Day 30
  Gingival Abrasion will be assessed with a 2-tone disclosing solution to help visualize abraded areas of the oral epithelium. Gingival tissues of each tooth will be divided into 3 areas on both the facial and lingual surfaces, as illustrated in Fig. 1: marginal (cervical free gingiva), interdental (papillary free gingiva) and mid-gingival (attached gingiva). If abrasion is present, the site will be recorded as small (≤2 mm), medium (3-5 mm) and large (>5 mm). If no abrasion is present, the site will be recorded as "0".

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Inc, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No